CLINICAL TRIAL: NCT06258590
Title: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) for the Treatment of Anxiety Comorbid With Autism Spectrum Disorder (ASD)
Brief Title: taVNS for Anxiety in ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00128238
Record Dates: First submitted 2024-01-09; First posted 2024-02-14 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Anxiety
Keywords: Brain stimulation; Transcutaneous auricular vagus nerve stimulation
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tVNS (Experimental): All patients will receive at-home Transcutaneous auricular vagus nerve stimulation (taVNS) and assess the impact on multiple behavioral outcomes associated with ASD and anxiety. This is an open-label trial.
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — Patients will receive non invasive vagus nerve stimulation via electrodes attached to the ear.

SUMMARY:
Investigators will recruit up to 10 patients with Anxiety comorbid with Autism Spectrum Disorder (ASD) from the outpatient clinics at MUSC. This pilot trial will be an open-label investigation of the safety and feasibility of transcutaneous auricular vagus nerve stimulation (taVNS) as a nonpharmacological wearable intervention used to manage anxiety and other neuropsychiatric symptoms at home, with patients/caretakers self-administering treatments. Each subject will undergo an initial in-person screening and be consented prior to participating in the study. This will be followed by an in-person training session with the subject (and caretaker if applicable), where they will learn how to self-administer taVNS and ask any pertinent questions. Participants will self-administer taVNS at home twice daily for 4 weeks. These treatments will not interfere with other aspects of their mental health care. Our investigators, over the prior 8 years, have demonstrated that taVNS is safe and feasible in the outpatient setting. Furthermore, investigators have recently demonstrated that taVNS is well tolerated and safely self-administered at home with remote monitoring. The investigators hypothesize that taVNS will be safe and feasible to administer at home in this new population. Results from this study may lead to further exploration of taVNS in this unique population.

DETAILED DESCRIPTION:
This is a research study to find out if anxiety in patients with autism spectrum disorder are affected by a form of ear stimulation called transcutaneous auricular vagus nerve stimulation, or taVNS. Participants will learn how to self-administer ear stimulation treatments at home before starting the study. Over the course of a month, participants will self-administer ear stimulation treatments twice a day for a month. Each treatment will last up to 60 minutes (1 hour) and there will be a break of at least 30 minutes in between treatments. The study team will ask participants to complete a group of questionnaires at the beginning and end of the study. There will also be a smaller number of questionnaires completed electronically on a weekly basis. The questionnaires will ask questions about mental health symptoms that subjects may or may not be experiencing, including questions about mood, anxiety, and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-17
* English speaking
* Prior diagnosis of ASD using autism diagnostic observation schedule (ADOS)
* Score >24 on SCARED
* IQ >70
* Have the capacity and ability to provide one's own assent, consent will be provided by legal guardian

Exclusion Criteria:

* Facial or ear pain or recent ear trauma.
* Metal implant devices in the head, heart or neck.
* History of brain surgery.
* History of myocardial infarction or arrhythmia, bradycardia.
* Acute exacerbation of a chronic respiratory disorder or acute COVID-related symptoms.
* Active GI symptoms with a history of diabetes mellitus or history of gastroparesis secondary to diabetes mellitus.
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Individuals with a reported history of psychosis or mania, or individuals who are actively manic or psychotic.
* Individuals who are catatonic or otherwise unable to participate in the informed consent process.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing adverse outcomes as measured by questionnaire | 4 weeks during trial with 30 day follow-up to assess adverse effects
  Assessing adverse outcomes via qualitative questionnaire asking participants about experiences during stimulation and any consequences after stimualtion

SECONDARY OUTCOMES:
Anxiety rating for participants using generalized anxiety disorder -child scale | Testing occurs prior to testing, at two weeks, and following the 4 week trial, along wioth a 30-day post trial follow-up
  Assessing the impact of stimulation on GAD-child scale, where lower numbers (0=none, 4=extreme) show improved anxiety
Empagthic abilities as measured by the Toronto Empathy Questionnaire | Testing occurs prior to testing, at two weeks, and following the 4 week trial, along wioth a 30-day post trial follow-up
  Assessing the participants change in the ability to identify the emotions of others using the TEQ, while a score of less than 45 indicating below average empathy levels, and a max score of 64

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT06258590/ICF_000.pdf